CLINICAL TRIAL: NCT03314766
Title: Evaluation of Long-Term Clinical Acceptability and Satisfaction With the IC-8 Intraocular Lens
Status: Completed | Type: Observational
Sponsor: AcuFocus, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IC-8 203-LTCA
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2018-07

CONDITIONS: Cataract; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- IC-8 IOL: Patients previously implanted with an IC-8 IOL contralaterally or bilaterally under the protocol ACU-P14-029
  Interventions: Device: IC-8 IOL

INTERVENTIONS:
Device: IC-8 IOL — Patients previously implanted with an IC-8 IOL contralaterally or bilaterally will be evaluated for their long-term visual functions and overall satisfaction at least 12 months post-implantation

SUMMARY:
The purpose of this study is to evaluate the long-term clinical acceptability and overall satisfaction with the IC-8 IOL at least 12 months post-IOL implantation.

DETAILED DESCRIPTION:
This will be a prospective, multi-center, non-interventional study in up to 80 patients previously implanted with an IC-8 IOL contralaterally or bilaterally under the protocol ACU-P14-029 at up to nine clinical sites within Europe.

The purpose of this study is to demonstrate the long-term clinical acceptability and overall satisfaction in patients implanted with the IC-8 IOL. The primary study endpoint is binocular target-corrected near visual acuity (TCNVA) of 20/32 or better in 85% or more patients at least 12 months post-implantation. The secondary study endpoint is overall satisfaction with postoperative vision in 85% or more patients reporting either satisfied or very satisfied at least 12 months post-implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients previously implanted contralaterally or bilaterally with the IC-8 IOL under the protocol ACU-P14-029 and have had the IOL implanted for a duration of at least 12 months and currently have the IC-8 IOL in the eye.
2. Availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures at the study visit.
3. Signed informed consent.

Exclusion Criteria:

1. Patients who have developed systemic or ocular pathology, not related to the IOL that affected their best corrected distance visual acuity to be 0.8 decimal or worse as determined by diagnostic testing or investigator's medical judgment. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for this study will be recruited from the clinical sites that participated in the prior open-label, multicenter study (protocol ACU-P14-029). Anticipated study sample size of no more than 80 patients should effectively demonstrate the long-term clinical acceptability of the IC-8 IOL implanted in aphakic patients.
  Patients will be screened for eligibility, and an informed consent will be obtained from those who meet the screening criteria and are interested in participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
TCNVA | 12 months
  Binocular target-corrected near visual acuity (TCNVA) of 20/32 or better in 85% or more patients.

SECONDARY OUTCOMES:
Overall Satisfaction | 12 months
  Overall satisfaction with postoperative vision at least 12 months post-operatively, with an outcome of objective of 85% or more being either very satisfied or satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Tarantino, OD, Study Director
Locations (7):
- Germany (2):
  - Augen Zentrum Nordwest, Ahaus
  - Universitats-Augenklinik, Department of Ophthalmology, Bochum
- Italy (2):
  - San Bassano Hospital, Bassano del Grappa
  - Centro Microchirurgia Ambulatoriale, Monza
- Ifocus Øyeklinikk, Haugesund, Norway
- Spain (2):
  - QVision (Unidad Oftalmología Hospital Virgen del Mar), Almería
  - Hospital Universitario Donostia, Servicio de Oftalmología, Donostia / San Sebastian

IPD SHARING:
Plan to Share IPD: No